CLINICAL TRIAL: NCT00265538
Title: Implementing Evidence-based Treatment of Hypertension
Brief Title: Implementing Evidence Based Treatment of Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IMV 04-066
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: Hypertension; Diuretics; Drug Therapy; Anti-Hypertensive Agents; Patient Intervention
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Pure Control Group) (No Intervention): Pure control (no intervention letter);
- Arm 2 (Contaminated Control Group) (No Intervention): Intervention control (patient does not receive intervention letter, but provider sees other patients who may bring in letter);
- Arm 3 (Intervention Group A) (Experimental): Intervention group A (the intervention is a letter only mailed to the subject); This intervention group receives an educational letter, which is the intervention. It is an educational intervention only.
  Interventions: Behavioral: Patient educational letter to engage provider in hypertension rx discussion
- Arm 4 (Intervention Group B) (Experimental): Intervention group B (intervention letter A + financial incentive for discussion w/ provider and 6 month copay reimbursement); This group receives the same educational intervention as Group A, but also receives the Financial incentive, which is an added intervention.
  Interventions: Behavioral: Patient educational letter to engage provider in hypertension rx discussion
- Arm 5 (Intervention Group C) (Experimental): Intervention group C (intervention letter A, financial incentive for discussion w/ provider + copay reimbursement, PLUS reminder phone call 1-3 days prior to primary care visit). This group receives the same intervention as Group B, but with the added intervention of a reminder phone call to test whether additional prompting is needed to make the intervention more effective.
  Interventions: Behavioral: Patient educational letter to engage provider in hypertension rx discussion; Behavioral: Financial incentive (Arms B and C) and health educator phone call (Arm C)

INTERVENTIONS:
Behavioral: Patient educational letter to engage provider in hypertension rx discussion — Patients will receive a customized/tailored letter (education) including most recent clinic blood pressure, current blood pressure medications and suggested htn medication(s). All the intervention arms (A, B and C) receive the letter.
  Arms: Arm 3 (Intervention Group A); Arm 4 (Intervention Group B); Arm 5 (Intervention Group C)
Behavioral: Financial incentive (Arms B and C) and health educator phone call (Arm C) — Patients may receive a financial incentive for discussing the intervention letter with their provider and 6 months copay reimbursement and/or the financial incentive discussion incentive, 6 months copay reimbursement as well as a phone call reminder 1-2 days prior to their primary care appt. The Financial incentive is part of both Arms B and C. The health educator phone call is only in Arm C.
  Arms: Arm 5 (Intervention Group C)

SUMMARY:
This study examines the use of patient initiated discussions of blood pressure medication in the primary care setting. Additionally, this study examines different levels of patient incentive(s) to initiate discussions with providers including information only, information plus a financial incentive and reimbursement for 6 months of copay, and information/monetary incentive plus a reminder call prior to the index visit. Patient opinions about doctor/patient relationships will be assessed. Provider attitudes and prescribing behaviors will be analyzed as well.

DETAILED DESCRIPTION:
Patients will be randomized to Pure control, intervention control, intervention group a, intervention group b or intervention group c. Pure control patients will not receive any study information about diuretics and their providers will not see any patients who receive our study intervention letter. Patients in the intervention control group will not receive the intervention but will see providers who have other patients in the intervention groups. Patients in intervention group a will receive a customized letter prior to their next primary care appointment with information regarding the patient's specific blood pressure, current blood pressure medication and recommendation for switching or adding a thiazide. Patients in group b will receive the customized intervention letter as well as a financial incentive for discussing the information with their provider and a copay reimbursement for 6 months if a prescription is written for a thiazide. Patients in group c will receive the intervention letter, financial discussion incentive, copay reimbursement as well as a phone call reminder 1-2 days prior to their primary care visit.

ELIGIBILITY:
Inclusion Criteria:

The eligible population includes patients less than 80 years of age enrolled in primary care clinics at the study sites that meet the following additional inclusion criteria:

* No active prescription for a thiazide diuretic (or a medication that combines a thiazide and another agent (e.g., hydrochlorothiazide and triamterene)
* Prior diagnosis of hypertension, as documented in VA outpatient administrative files
* Two or more visits to a primary care clinic in the prior 12 months;
* Blood pressure above treatment goal at the two most recent VA outpatient clinic visits Above goal is defined as a systolic pressure >140 mmHg or diastolic pressure >90 mmHg. For diabetics above goal is defined as systolic pressure >130 mmHg or diastolic pressure >80 mmHg
* Blood pressure at goal (as defined above) during one of the last two outpatient clinic visits, but the patient is receiving a prescription for a calcium channel blocker (CCB)

Exclusion Criteria:

Patients meeting the above inclusion criteria will be excluded for the following reasons:

* Documented allergy to thiazides or to sulfa agents
* Previously documented intolerance or adverse drug reaction to thiazide diuretics
* Active prescription for a loop diuretic agent (e.g. furosemide)
* Renal insufficiency, defined by a glomerular filtration rate less than 30 ml/min
* No serum creatinine in the past year (to permit calculation of a creatinine clearance)
* Prior history of hypokalemia or serum potassium less than 3.5 meq/l in the prior year
* Diagnosis of gout or active prescription for allopurinol
* Congestive heart failure (CHF) due to systolic dysfunction with a documented left ventricular ejection fraction < 35% by echocardiography, nuclear medicine study, or ventriculography
* Residence in a long-term care facility
* No telephone for follow-up calls
* Life-expectancy < 6 months
* Inability to give informed consent or impaired cognitive function (defined as > 4 errors on the 10-item Pfeiffer Portable Mental Status Questionnaire82, administered during study intake)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2006-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Kaboli, MD MS, Principal Investigator — VA Medical Center, Iowa City
Locations (2):
- United States (2):
  - VA Medical Center, Iowa City, Iowa City, Iowa
  - Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota

REFERENCES:
- [Result] Kaboli PJ, Shivapour DM, Henderson MS, Barnett MJ, Ishani A, Carter BL. Patient and provider perceptions of hypertension treatment: do they agree? J Clin Hypertens (Greenwich). 2007 Jun;9(6):416-23. doi: 10.1111/j.1524-6175.2007.06492.x. PMID 17541326
- [Result] Pilling SA, Williams MB, Brackett RH, Gourley R, Weg MW, Christensen AJ, Kaboli PJ, Reisinger HS. Part I, patient perspective: activating patients to engage their providers in the use of evidence-based medicine: a qualitative evaluation of the VA Project to Implement Diuretics (VAPID). Implement Sci. 2010 Mar 18;5:23. doi: 10.1186/1748-5908-5-23. PMID 20298563
- [Result] Buzza CD, Williams MB, Vander Weg MW, Christensen AJ, Kaboli PJ, Reisinger HS. Part II, provider perspectives: should patients be activated to request evidence-based medicine? A qualitative study of the VA project to implement diuretics (VAPID). Implement Sci. 2010 Mar 18;5:24. doi: 10.1186/1748-5908-5-24. PMID 20298564
- [Result] Sutton E, Wilson H, Kaboli PJ, Carter BL. Why physicians do not prescribe a thiazide diuretic. J Clin Hypertens (Greenwich). 2010 Jul 1;12(7):502-7. doi: 10.1111/j.1751-7176.2010.00299.x. PMID 20629812
- [Result] Reisinger HS, Brackett RH, Buzza CD, Paez MB, Gourley R, Weg MW, Christensen AJ, Kaboli PJ. "All the money in the world ..." patient perspectives regarding the influence of financial incentives. Health Serv Res. 2011 Dec;46(6pt1):1986-2004. doi: 10.1111/j.1475-6773.2011.01287.x. Epub 2011 Jun 20. PMID 21689098
- [Result] Kaboli PJ, Baldwin AS, Henderson MS, Ishani A, Cvengros JA, Christensen AJ. Measuring preferred role orientations for patients and providers in veterans administration and university general medicine clinics. Patient. 2009 Mar 1;2(1):33-8. doi: 10.2165/01312067-200902010-00004. PMID 22273057
- [Result] Lund BC, Charlton ME, Steinman MA, Kaboli PJ. Regional differences in prescribing quality among elder veterans and the impact of rural residence. J Rural Health. 2013 Spring;29(2):172-9. doi: 10.1111/j.1748-0361.2012.00428.x. Epub 2012 Aug 27. PMID 23551647
- [Derived] Howren MB, Vander Weg MW, Christensen AJ, Kaboli PJ. Association of patient preferences on medication discussion in hypertension: Results from a randomized clinical trial. Soc Sci Med. 2020 Oct;262:113244. doi: 10.1016/j.socscimed.2020.113244. Epub 2020 Jul 29. PMID 32750626
- [Derived] Kaboli PJ, Howren MB, Ishani A, Carter B, Christensen AJ, Vander Weg MW. Efficacy of Patient Activation Interventions With or Without Financial Incentives to Promote Prescribing of Thiazides and Hypertension Control: A Randomized Clinical Trial. JAMA Netw Open. 2018 Dec 7;1(8):e185017. doi: 10.1001/jamanetworkopen.2018.5017. PMID 30646291

RESULTS

PARTICIPANT FLOW:
Recruitment Details: An intervention study was implemented. Both the Iowa City VA and associated outpatient clinics as well as the Minneapolis VA and associated clinics were sites chosen for this intervention study. Subjects with a diagnosis of uncontrolled Hypertension or Hypertension controlled by a CCB were recruited.
Pre-assignment Details: 61,019 potential subjects from the 13 clinics were screened using an automated protocol to identify 2,910 potentially eligible subjects
Groups:
- Intervention Group A: Group a (intervention letter only): Patients will receive a customized/tailored letter including most recent clinic blood pressure, current blood pressure medications, and suggested blood pressure medication(s). The letter also encouraged the patient to discuss their blood pressure treatment with their provider.
- Intervention Group B: Group B: intervention letter from Group A + $20 financial incentive for discussion with the provider and 6 month copay reimbursement if the patient has a copay.
- Intervention Group C: Group C: Intervention letter from Group A + financial incentive from Group B + health educator phone call. The phone call 1-2 days prior to their primary care appointment encouraged them to talk with their provider about their blood pressure treatment.
- Control Group: The control group received usual care. They were given informed consent that they could either be in the intervention or control groups.
Period: Overall Study
Arm/Group | Intervention Group A | Intervention Group B | Intervention Group C | Control Group
Started | 196 | 170 | 182 | 286
Completed | 186 | 161 | 171 | 267
Not Completed | 10 | 9 | 11 | 19

BASELINE CHARACTERISTICS:
Population: Baseline data were only collected as combined control and intervention groups and it is not possible to separate by the 3 arms of the intervention for separate analysis. Because of randomization, the difference in baseline characteristics should not be meaningfully different.
Groups:
- Control Group: No intervention (usual care)
- Combined Intervention Groups: Patient Intervention Arms: Group A (intervention letter only); Group B (intervention, + financial incentive for discussion w/ provider and 6 month copay reimbursement); Group C (intervention letter, financial incentive for discussion w/ provider + copay reimbursement, plus reminder phone call 1-3 days prior to primary care visit)
- Total: Total of all reporting groups
Arm/Group | Control Group | Combined Intervention Groups | Total
Number analyzed (Participants) | 286 | 548 | 834
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (9.2) | 62.9 (8.8) | 63.1 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 13
  Male | 282 | 539 | 821
Region of Enrollment [Number; unit: participants]
  United States | 286 | 548 | 834

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients Taking Thiazide Diuretics and at BP Goal at Index Visit and 6 Months
Description: Reported in 2 sub-groups: Subgroup 1 not at BP goal; Subgroup 2 at BP goal but taking a calcium channel blocker (see pre-specified sub group analysis below).
Time Frame: index visit and 6 months
Population: Total number of patients prescribed a thiazide at time of enrollment (index visit).
Measure: Count of Participants; unit: Participants
Groups:
- Intervention Group A: Group A (intervention letter only)
- Intervention Group B: Intervention Letter + financial incentive
- Intervention Group C: Intervention letter + financial incentive + phone call
- Control Group: Usual care
Arm/Group | Intervention Group A | Intervention Group B | Intervention Group C | Control Group
Number analyzed (Participants) | 143 | 128 | 131 | 196
Participants
  Taking Thiazide at Index (baseline) visit | 35 | 33 | 43 | 19
  At BP goal at Index (baseline) visit | 29 | 31 | 33 | 45
  Taking Thiazide at 6 months | 31 | 28 | 37 | 31
  At BP goal at 6 months | 38 | 39 | 40 | 48

2. Other Pre Specified Outcome: Percent of Patients Taking a Thiazide at Baseline (Subgroup 2 at BP Goal and Taking a Calcium Channel Blocker)
Description: This was a pre-specified sub-group of patients already at their blood pressure goal, so the primary outcome was taking a thiazide at baseline (index visit).
Time Frame: At index visit
Population: The number of participants analyzed represents the number of participants with available data at each time point. This was a pre-specified sub-group and there for did not have the entire study population represented.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Group A | Intervention Group B | Intervention Group C | Control Group
Number analyzed (Participants) | 53 | 42 | 51 | 90
Participants | 5 | 11 | 16 | 1

ADVERSE EVENTS:
Description: There were not any reported Adverse Events, so there is not separate reporting of events, because there were no events. The numerator for all is zero.
  Because there were no events, the denominator was combined into all the Control Patients and all the Intervention Patients. It is thus not possible to separate them since there were no events.
Groups:
- Combined Intervention Groups: Patient Intervention Arms: Group A (intervention letter only); Group B (intervention, + financial incentive for discussion w/ provider and 6 month copay reimbursement); Group C (intervention letter, financial incentive for discussion w/ provider + copay reimbursement, plus reminder phone call 1-3 days prior to primary care visit)blood pressure, current blood pressure medications and suggested htn medication(s)
Arm/Group | Control Group | Combined Intervention Groups
All-Cause Mortality (participants affected / at risk) | 0/286 | 0/548
Serious Adverse Events (participants affected / at risk) | 0/286 | 0/548
Other Adverse Events (participants affected / at risk) | 0/286 | 0/548
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=286) | Combined Intervention Groups (N=548)
(Blood and lymphatic system disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No